CLINICAL TRIAL: NCT00819858
Title: The Effectiveness of Ready to Use Therapeutic Food (RUTF) in Catch up Growth in Children After an Episode of P. Falciparum Malaria
Brief Title: Effect of Ready to Use Therapeutic Food (RUTF) Supplement After an Episode of Malaria Falciparum on Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Saskia van der Kam, Ir, Medecins Sans Frontieres, Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSF-nutcon01
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Weight Loss; Weight Gain; Convalescence; Malaria
Keywords: weight loss; weight gain; malnutrition; convalescence; malaria; RUTF; RUF; supplementation; nutrition
MeSH Terms: conditions — Weight Loss; Weight Gain; Convalescence; Malaria; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RUTF (Experimental): RUTF supplement (Plumpynut®) of 500 kcal/day for 2 weeks
  Interventions: Dietary Supplement: RUTF (Plumpynut®)
- control (No Intervention): no supplement given

INTERVENTIONS:
Dietary Supplement: RUTF (Plumpynut®) — Intervention group receives 500 kcal/day of RUTF for 2 weeks Control group receives no food supplement
  Other Names: RUTF; Ready to use Therapeutic Food; RUF; Lipid based food supplement
  Arms: RUTF

SUMMARY:
The primary objective of this study is to determine to what extent provision with RUTF will promote catch up growth in children following an acute uncomplicated episode of P. falciparum malaria.

DETAILED DESCRIPTION:
Anorexia due to infection might lead to weight loss. In many settings total recovery is problematic what might result in a permanent lower weight. A short period high quality food supplementation could improve weight gain after an infection.

Children aged 6-59 months presenting with malaria caused by P. falciparum who are provided with a RUTF supplement (Plumpynut®) of 500 kcal/day for 2 weeks will show significantly better catch up growth compared to a similar patient group not provided with RUTF (at 2 weeks and 4 weeks post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 59 months, and
* Positive rapid diagnostic test (Paracheck®) and
* Thick smear showing infection with P. falciparum and
* Informed consent from parents or guardian aged at least 18 years.

Exclusion Criteria:

* Children who are exclusively breast fed or
* Children who are severely malnourished (MUAC <110 mm and/or bilateral oedema, or WHO weight-for-Height criteria <3 Z-scores) or
* Presence of general danger signs or signs of severe malaria as defined by the WHO criteria, or
* Known history of allergy to malaria drugs, or
* Having a sibling enrolled in the study.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
weight gain | 14 days

SECONDARY OUTCOMES:
weight gain | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Saskia van der Kam, Ir, Principal Investigator — nutrition expert MSF
Locations (1):
- Central Hospital, Dubie, Katanga, Republic of the Congo

REFERENCES:
- [Derived] van der Kam S, Swarthout T, Niragira O, Froud A, Sompwe EM, Mills C, Roll S, Tinnemann P, Shanks L. Ready-to-use therapeutic food for catch-up growth in children after an episode of Plasmodium falciparum malaria: an open randomised controlled trial. PLoS One. 2012;7(4):e35006. doi: 10.1371/journal.pone.0035006. Epub 2012 Apr 25. PMID 22558108